CLINICAL TRIAL: NCT03237871
Title: The Engaging Microenterprise for Resource Generation and Health Empowerment (EMERGE) Project: Feasibility of Assessing Economic and Sexual Risk Behaviors Using Text Messages in Homeless Young Adults
Brief Title: The EMERGE Project: Feasibility of Assessing Economic and Sexual Risk Behaviors Using Text Messages in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB0007563; K01MH107310 (NIH)
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey and informational text messages (Experimental): Text-message survey and informational text messages
  Interventions: Behavioral: Text-message survey and informational text messages

INTERVENTIONS:
Behavioral: Text-message survey and informational text messages — Participants will complete a text-messaged survey each week for 5 weeks assessing economic and sexual risk behaviors. Participants will also receive 3 informational text messages each week for 5 weeks on HIV prevention and economic empowerment.

SUMMARY:
As part of the development of the Engaging Microenterprise for Resource Generation and Health Empowerment (EMERGE) Project, the study team will conduct a single-group study to examine the feasibility of assessing economic and sexual risk behaviors using text messages. The team will enroll approximately 20 young adults, aged 18 to 24, who are African-American, homeless, out-of-school, and un/under-employed. Participants will complete a text-messaged survey each week for 5 weeks. The study team will collect information about the number of participants who respond to the weekly survey, the number of questions to which they respond in each survey, and the number of hours from sending a survey to participants to receiving their response. As an exploratory aim, participants will also receive 3 informational text messages each week for 5 weeks on HIV prevention and economic empowerment. The study team will obtain qualitative feedback from participants regarding text messages they most and least liked. The survey is not designed to evaluate the effectiveness of the text message intervention.

DETAILED DESCRIPTION:
As part of the development of the Engaging Microenterprise for Resource Generation and Health Empowerment (EMERGE) Project, the study team will conduct a single-group study to examine the feasibility of assessing economic and sexual risk behaviors using text messages. The study team will enroll approximately 20 young adults, aged 18 to 24, who are African-American, homeless, out-of-school, and un/under-employed. Participants will complete a text-messaged survey each week for 5 weeks. The study team will collect information about the number of participants who respond to the weekly survey, the number of questions to which they respond in each survey, and the number of hours from sending a survey to participants to receiving their response. As an exploratory aim, participants will also receive 3 informational text messages each week for 5 weeks on HIV prevention and economic empowerment. The study team will obtain qualitative feedback from participants regarding text messages they most and least liked. The survey is not designed to evaluate the effectiveness of the text message intervention. The single-group study is anticipated to start in August 2017.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be included in the study if, at the time of enrollment, they are:
* African American
* Aged 18-24
* Living in Baltimore City
* Experiencing homelessness in the past 12 months
* Employed fewer than 10 hours per week
* Not enrolled in school
* Ownership of a mobile phone with text-messaging capacity
* Reporting at least one episode of unprotected sex in prior 6 months or one other personal or sexual partner HIV risk factor within prior 6 months (STI diagnosis, sex while high or drunk, sex exchange, illicit drug use, alcohol dependence).

Exclusion Criteria:

* Aged 17 or younger.
* Older than 24 years
* Unwilling to provide consent for study participation

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Jennings, PhD MHS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol
Time Frame: De-identified individual patient data (IPD) that under results in a publication will become available 12 months after publication and will be available for 24 months.
Access Criteria: Sponsor approval for data sharing will be sought. Only bona fide research groups are eligible to access data as evidenced via curriculum vitae (CV) and the involvement of a qualified statistician or qualitative research scientist. Data access requests should be made via email application to the principal investigator detailing the specific requirements and the proposed research and publication plan. Data access requests will be reviewed against specific criteria by the data custodians. Decisions about requests will be made promptly and no more than 3 months after receipt of request.

REFERENCES:
- [Derived] Jennings Mayo-Wilson L, Glass NE, Labrique A, Davoust M, Ssewamala FM, Linnemayr S, Johnson MW. Feasibility of Assessing Economic and Sexual Risk Behaviors Using Text Message Surveys in African-American Young Adults Experiencing Homelessness and Unemployment: Single-Group Study. JMIR Form Res. 2020 Jul 17;4(7):e14833. doi: 10.2196/14833. PMID 32706656

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Survey and Informational Text Messages
Started | 17
Completed | 11
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Number of participants enrolled in the study
Arm/Group | Survey and Informational Text Messages
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Age] | 21.2 [18 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Recruited from community organization [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Respond to the Survey in Week 1
Description: Number of enrolled participants who respond to the survey in Week 1. Measure type 'number' was used for small sample size and as described in the original registration protocol.
Time Frame: Week 1
Population: Number of participants enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Survey and Informational Text Messages
Number analyzed (Participants) | 17
Participants | 7

2. Primary Outcome: Mean Number of Questions to Which Participant Respond in Each Survey in Week 1
Description: Mean number of questions to which enrolled participant respond in each survey in Week 1.
Time Frame: Week 1
Population: Mean number of participants enrolled in the study who responded to the survey in week 1
Measure: Mean (Standard Deviation); unit: Mean number of responded questions
Arm/Group | Survey and Informational Text Messages
Number analyzed (Participants) | 7
Mean number of responded questions | 10.1 (5.2)

3. Primary Outcome: Mean Number of Hours From Sending a Survey to Participants to Receiving Their Response in Week 1
Description: Mean number of hours from sending a survey to enrolled participants to receiving their response in Week 1.
Time Frame: Week 1
Population: Mean number of participants enrolled in the study who responded to the survey in week 1
Measure: Mean (Standard Deviation); unit: Mean number of hours
Arm/Group | Survey and Informational Text Messages
Number analyzed (Participants) | 7
Mean number of hours | 1.7 (2.2)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Survey and Informational Text Messages
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT03237871/Prot_SAP_000.pdf